CLINICAL TRIAL: NCT02637219
Title: Innate Immune Response in COPD
Status: Completed | Type: Observational
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: University of Washington (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Vincent S. Fan, Associate Professor, VA Puget Sound Health Care System
Other Study IDs: 01439
Record Dates: First submitted 2015-12-03; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Immunity, Innate; Inflammation; Bronchitis, Chronic; Toll-Like Receptors
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the response of the immune system to bacterial components differs between patients with severe COPD compared to those with less severe COPD.

DETAILED DESCRIPTION:
The airways of COPD patients are often colonized with bacteria leading to increased airway inflammation. This study sought to determine whether systemic cytokine responses to microbial pathogen-associated molecular patterns (PAMPs) are increased among subjects with severe COPD.

In an observational cross-sectional study of COPD subjects, PAMP-induced cytokine responses were measured in whole blood ex vivo. We used PAMPs derived from microbial products recognized by TLR 1, 2, 4, 5, 6, 7, and 8. Patterns of cytokine response to PAMPs were assessed using hierarchical clustering. One-sided t-tests were used to compare PAMP-induced cytokine levels in blood from patients with and without severe COPD, and for subjects with and without chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

* post-bronchodilator FEV1/FVC <0.7
* FEV1 < 80%
* > 10 pack-years tobacco smoking
* no respiratory illnesses or prednisone or antibiotics in the last 4 weeks

Exclusion Criteria:

* Primary diagnosis of asthma
* > 15% change in FEV1
* Chronic inflammatory or infectious disease
* Cancer
* Autoimmune disease
* Chronic renal failure with a creatinine > 1.5
* Chronic liver disease
* Chronic antibiotic use

Note: Due to difficulty recruiting patients after 6 participants were enrolled, the exclusion criteria were modified to allow patients with > 15% change in FEV1. The exclusion criteria were also changed to allow chronic renal failure not requiring dialysis, and non-metastatic cancer provided there was no diagnosis of lung cancer.

Ages: 50 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical history of COPD recruited from a pulmonary subspecialty clinic at an academic medical center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Cytokine production (TNF-alpha, IL-6, IL-8, IL-10, IL-1RA, G-CSF, IL-1B, MCP-1). | This is a cross-sectional study with no follow-up period. Therefore the study outcomes were measured at the baseline visit (Time = day 0)
  A whole blood stimulation assay was performed on blood samples from study participants. The whole blood was stimulated using several pathogen-associated molecular patterns that were agonists to seven different TLR receptors: 1) Pam3SCK4, 2) Zymosan, 3) FSL-1, 4) LPS, 5) flagellin, 6) R848. After stimulation with the PAMP, the cytokine levels (TNF-alpha, IL-6, IL-8, IL-10, IL-1RA, G-CSF, IL-1B, and MCP-1) were measured and the cytokine level results are in picograms per liter. Note, there is no treatment in this observational non-interventional trial. Therefore the multiple cytokine levels for each patient will not be aggregated or summarized into one measure. This study was a small pilot study and the results are exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Fan, MD MPH, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States